CLINICAL TRIAL: NCT04429555
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy, Safety, Tolerability, Biomarkers and Pharmacokinetics of Ibudilast (MN-166) in COVID-19 Subjects at Risk for Developing Acute Respiratory Distress Syndrome
Brief Title: Efficacy, Safety, Tolerability, and Biomarkers of Ibudilast (MN-166) in Patients Hospitalized With COVID-19 at Risk for ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MN-166-COVID-19-201
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pneumonia, Viral
Keywords: COVID-19; Acute respiratory distress syndrome; Pneumonia
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Respiratory Distress Syndrome; Pneumonia | interventions — ibudilast

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Experimental)
  Interventions: Drug: Ibudilast
- Placebo Treatment Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibudilast — 50 mg (5 x 10 mg capsules) twice daily for 7 days
  Other Names: MN-166
  Arms: Active Treatment Group
Drug: Placebo — 0 mg (5 matching capsules) twice daily for 7 days
  Arms: Placebo Treatment Group

SUMMARY:
The goal of this study is to evaluate the effects of Ibudilast (MN-166) versus placebo in hospitalized patients infected with COVID-19 at risk for developing acute respiratory distress syndrome (ARDS) receiving standard of care (including anticoagulation therapy) by measuring the following outcomes: 1) the need for oxygen therapy at Days 7, 14, and 28, 2) clinical status as measured by the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale at Days 7, 14, and 28, and 3) safety (as measured by incidence of adverse events and clinical laboratory findings) and tolerability of Ibudilast.

DETAILED DESCRIPTION:
This is a randomized (1:1) double-blind, placebo-controlled, parallel-group study evaluating the efficacy of Ibudilast to prevent ARDS in hospitalized patients infected with COVID-19 who are at risk for developing ARDS. The study will consist of a Screening Phase, Double-Blind Treatment Phase, and Follow-up Phase. Following the Screening Phase, if the participant meets eligibility criteria, they will be randomly assigned to Ibudilast or matching placebo. Participants will receive Ibudilast 100 mg/d (50 mg twice a day) or placebo every day for 7 days. Upon completion of the 7-day Treatment Phase, subject will be followed-up at Day 14 and at Day 28. Participants discharged prior to Day 7 will be given the remainder of their study medication (Ibudilast or placebo) to be taken at home twice daily until Day 7 and will be given a pulse oximeter to measure their oxygen levels once daily until Day 14.

The following screening assessments will be performed upon signing the Informed Consent Form (ICF): inclusion/exclusion criteria review, physical exam, vital signs and oxygen use, clinical status using the NIAID ordinal scale, 12-lead ECG, blood collection for plasma biomarkers. A complete blood count (CBC), comprehensive metabolic panel (CMP), D-dimer and coagulation tests will also be drawn. A serum pregnancy test will be given to pre-menopausal female participants. Concomitant medications taken within the last 7 days prior to study drug administration will be recorded.

During the Treatment Phase, hospitalized participants will be treated with Ibudilast or placebo for a 7-day period plus standard of care and anticoagulation therapy. During the Treatment Phase, participants will undergo study-related procedures including physical exam, ECG, oxygen use assessment, biomarkers and pharmacokinetic sample draws, CBC, CMP, D-dimer blood collection, clinical status using the NIAID scale, and information on adverse events and concomitant medications will be recorded.

On Study Day 14, conduct physical examination, clinical status, vital signs and oxygen use, ECG, CBC, CMP, D-dimer, and coagulation tests, biomarkers, AE and concomitant medications review. On Day 28, participant's clinical status and survival status will be recorded.

If the participant is discharged before Day 7, they will be given the remainder of their study drug to take at home for up to 7 days, and the Sponsor will supply a pulse oximeter to participants to measure their oxygen levels once daily until Day 14.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed with WHO criteria (including a positive PCR of any specimen, e.g., blood, respiratory, stool, urine, or any other body fluid)
* Chest imaging (radiograph, computerized tomography (CT) scan or lung ultrasound) with abnormalities consistent with COVID-19 pneumonia
* Oxygen saturation (SpO2) ≤92% on room air (RA), respiratory rate ≥24 breaths per min on RA, and/or requirement for supplemental oxygen
* At least 1 risk factor which may put patient at higher risk for more severe illness from COVID-19: Age > 65, underlying serious heart disease, chronic lung disease, moderate to severe asthma, body mass index of ≥40, or diabetes

Exclusion Criteria:

* Suspected active bacterial, fungal, viral, or other cause of respiratory failure other than COVID-19
* Subject is already intubated and on ventilator support
* Known or suspected immunosuppression with immunosuppressant medications or chemotherapeutic agents
* Patient is receiving dialysis treatment
* On a home ventilator support or continuous domiciliary oxygen therapy for baseline lung disease
* Active tuberculosis infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Matsuda, MD PhD MPH, Study Chair — Medicinova Inc
Locations (2):
- United States (2):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * Full Analysis Set (FAS) will include all participants randomly assigned to Ibudilast or placebo.
  * Safety Analysis Set (SAS) will include all randomized subjects who received at least one dose of study drug and had at least one post-dose safety assessment.
  * Per Protocol Analysis (PP): will consist of the FAS subjects excluding those with major protocol violations.
  In this clinical trial, FAS, SAS, and PP analysis sets included all participants.
Groups:
- Ibudilast (MN-166): 50 mg (10 mg strength): 5 capsules taken by mouth twice daily for 7 days.
- Placebo: 0 mg: 5 capsules taken by mouth twice daily for 7 days.
Period: Overall Study
Arm/Group | Ibudilast (MN-166) | Placebo
Started | 17 | 17
Completed | 15 | 15
Not Completed | 2 | 2
Not completed — Death | 0 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibudilast (MN-166) | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.71 (11.32) | 61.06 (12.16) | 59.88 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 10 | 13 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Respiratory Failure at Day 7
Description: Participants were considered "responders" if they did not meet the need for supplemental oxygen requirements (invasive mechanical ventilation, non-invasive ventilation, high-flow oxygen, or ECMO, CPAP, BiPAP, nasal cannula) at the end of the 7-day double-blind treatment.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast (MN-166) | Placebo
Number analyzed (Participants) | 17 | 17
Participants | 12 | 6

2. Primary Outcome: Number of Participants With at Least a 1-point Improvement in Clinical Status on Day 7
Description: Number (percentage) of participants with at least a 1-point improvement in clinical status on Day 7. Clinical status is measured by the National Institute of Allergy and Infectious Disease (NIAID) 8-Point Ordinal Scale: 1=Not hospitalized, no limitations on activities; 2=Not hospitalized, limitation on activities and/or requiring home oxygen; 3=Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 4=Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise) 5=Hospitalized, Hospitalized, requiring supplemental oxygen; 6=Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7=Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8=Death.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast (MN-166) | Placebo
Number analyzed (Participants) | 17 | 17
Participants | 12 | 8

3. Secondary Outcome: Number of Participants Receiving Mechanical Ventilation or Intubation
Description: Number (percentage) of participants receiving mechanical ventilation or intubation after starting study drug.
Time Frame: Days 7, 14, and 28
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast (MN-166) | Placebo
Number analyzed (Participants) | 17 | 17
Participants
  Day 7 | 1 | 3
  Day 14 | 1 | 2
  Day 28 | 1 | 1

4. Secondary Outcome: All-cause Mortality
Description: Number of reported participant deaths
Time Frame: Day 1 to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast (MN-166) | Placebo
Number analyzed (Participants) | 17 | 17
Participants | 0 | 2

5. Secondary Outcome: Number of Participants Discharged From Hospital at Days 7, 14, and 28
Description: Number (percentage) of participants discharged from hospital at Days 7, 14, and 28
Time Frame: Days 7, 14, and 28
Measure: Count of Participants; unit: Participants
Arm/Group | Ibudilast (MN-166) | Placebo
Number analyzed (Participants) | 17 | 17
Participants
  Day 7 | 11 | 5
  Day 14 | 13 | 11
  Day 28 | 13 | 14

ADVERSE EVENTS:
Time Frame: Adverse events occurring from the time of the first dose through 7 days after the last dose of MN-166 were recorded.
Groups:
- MN-166 (Ibudilast): 50 mg (10 mg strength): 5 capsules taken by mouth twice daily for 7 days.
Arm/Group | MN-166 (Ibudilast) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 5/17 | 14/17
Other Adverse Events (participants affected / at risk) | 13/17 | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MN-166 (Ibudilast) (N=17) | Placebo (N=17)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — Constipation
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Renal and urinary disorders) | 2 (3) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MN-166 (Ibudilast) (N=17) | Placebo (N=27)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0/17 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 3/17 (3)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1/17 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1/17 (1)
Bradycardia (Cardiac disorders) | 7 (7) | 3/17 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1/17 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0/17 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1/17 (1)
Glucose tolerance impaired (Endocrine disorders) | 0 (0) | 1/17 (1)
Hyperglycaemia (Endocrine disorders) | 0 (0) | 3/17 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2/17 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0/17 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1/17 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0/17 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0/17 (0)
Asthenia (General disorders) | 0 (0) | 1/17 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1/17 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0/17 (0)
Sepsis (Infections and infestations) | 1 (1) | 1/17 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0/17 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0/17 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1/17 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1/17 (1)
Transaminases increased (Investigations) | 1 (1) | 4/17 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1/17 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1/17 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1/17 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1/17 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1/17 (1)
Headache (Nervous system disorders) | 1 (1) | 2/17 (2)
Insomnia (Nervous system disorders) | 1 (1) | 1/17 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0/17 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0/17 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0/17 (0)
Depression (Psychiatric disorders) | 1 (1) | 0/17 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0/17 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0/17 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0/17 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2/17 (2)
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1/17 (1)
Hypotension (Vascular disorders) | 0 (0) | 2/17 (2)
Tongue haemorrhage (Vascular disorders) | 0 (0) | 1/17 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04429555/Prot_SAP_ICF_000.pdf